CLINICAL TRIAL: NCT00872157
Title: A Limited, First-in-Man, Phase IB Evaluation of BMTP-11 in Patients With Castrate-Resistant Prostate Cancer With High-Volume Osseous Metastases and no Standard Treatment Options
Brief Title: BMTP-11 in Patients With Castrate-Resistant Prostate Cancer With Bone Mets
Status: Completed | Phase: Phase 1 | Type: Interventional
Sponsor: M.D. Anderson Cancer Center (Other)
Responsible Party: Sponsor
Allocation: Not Applicable | Model: Single Group | Masking: None | Purpose: Treatment
Other Study IDs: 2008-0395; NCI-2012-01626 (Registry Identifier: NCI CTRP)
Record Dates: First submitted 2009-03-30; First posted 2009-03-31 (Estimated); Last update posted 2015-10-23 (Estimated); Status verified 2015-10

CONDITIONS: Prostate Cancer
Keywords: Castrate-Resistant Prostate Cancer; Prostate; High-Volume Osseous Metastases; BMTP-11; Prostate State Antigen; PSA
MeSH Terms: conditions — Prostatic Neoplasms | interventions — bone metastasis-targeting peptidomimetic-11

STUDY DESIGN:
Oversight: Data Monitoring Committee: No

ARMS (1):
- BMTP-11 (Experimental): Starting Dose of 6 mg/m2 by vein over 2 hours on Days 1, 8, 15, and 22.
  Interventions: Drug: BMTP-11

INTERVENTIONS:
Drug: BMTP-11 — Starting Dose of 6 mg/m2 by vein over 2 hours on Days 1, 8, 15, and 22.

SUMMARY:
The goal of this clinical research study is find the highest tolerable dose of BMTP-11 when given to patients with prostate cancer that has spread. The safety of this drug will also be studied.

DETAILED DESCRIPTION:
The Study Drug:

BMTP-11 is designed to use a protein to bind to cancer cells, move into the cancer cells, and cause the cancer cells to die. This is the first study using BMTP-11 in humans.

Study Groups:

If you are found to be eligible to take part in this study, you will be assigned to a dose level of BMTP-11 based on when you joined this study. Up to 2 dose levels of BMTP-11 will be tested. Three (3) participants will be enrolled at each dose level. The first group of participants will receive the lowest dose level. Each new group will receive a higher dose than the group before it, if no intolerable side effects were seen. This will continue until the highest tolerable dose of BMTP-11 is found.

Study Drug Administration:

On Days 1, 8, 15, and 22 of each cycle, you will receive BMTP-11 though a needle into your vein over 2 hours.

Before each dose of BMTP-11, you will receive saline (salt water) by vein for over 2 hours.

Study Visits:

On Days 7 and 14 of Cycles 1 and 2, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs, height, and weight.
* Your performance status will be recorded.
* You will be asked about any drugs you may be taking and if you have experienced any side effects.
* Blood (about 3 teaspoons) will be collected for routine tests. A portion of this blood will also be used to check your heart health.
* Urine will be collected over 24 hours to test your kidney function.

On Day 21 of Cycles 1 and 2, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs, height, and weight.
* Your performance status will be recorded.
* You will be asked about any drugs you may be taking and if you have experienced any side effects.
* Blood (about 3 teaspoons) will be collected for routine tests. A portion of this blood will also be used to check your heart health.
* Blood (about 1 teaspoon) will be drawn to measure your prostatic specific antigen (PSA) and testosterone levels.
* Urine will be collected over 24 hours to test your kidney function.

On Day 1 of Cycle 2, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs, height, and weight.
* Your performance status will be recorded.
* You will be asked about any drugs you may be taking and if you have experienced any side effects.
* Blood (about 3 teaspoons) will be collected for routine tests. A portion of this blood will also be used to check your heart health.
* Blood (about 1 teaspoon) will be drawn to measure your PSA and testosterone levels.

Length of Study:

You will be on active study for up to 9 weeks. You will be taken off study if you experience intolerable side effects or the disease gets worse. Please note that even if the treatment has a beneficial effect on the cancer, the treatment cannot be continued for more than two cycles due to the very limited supply of drug available.

End-of-Study Visit:

Between 4 and 6 weeks after the last dose of study drug, you will have an end-of-study visit. At this visit, the following tests and procedures will be performed:

* You will have a physical exam, including measurement of your vital signs, height, and weight.
* Your performance status will be recorded.
* You will be asked about any drugs you may be taking and if you have experienced any side effects.
* Blood (about 3-4 teaspoons) and urine will be collected for routine tests. This routine blood draw will include measurement of your PSA and testosterone levels. A part of this blood will also be used to see if your immune system reacted to BMTP-11 by forming an antibody and to assess your heart's health.
* Urine will be collected for 24 hours to test for protein in your urine.
* You will have CT or MRI scans of your abdomen and pelvis to check the status of the disease.
* You will have a chest x-ray.
* You will have a bone scan to check the status of the disease.

Follow-Up:

At 3, 6, and 9 months after the last dose of study drug, you will be called or e-mailed and asked how you are doing. This will only take a few minutes. You will be required to have blood drawn (about 1 teaspoon) for routine testing. This can be done at your local doctor's office and results faxed to MD Anderson Cancer Center (MDACC).

This is an investigational study. BMTP-11 is not FDA approved or commercially available. At this time, BMTP-11 is only being used in research.

Up to 22 patients will take part in this study. All will be enrolled at M. D. Anderson.

ELIGIBILITY:
Inclusion Criteria:

1. Have histologically confirmed adenocarcinoma of the prostate, with clinically significant bone metastases exhibiting castrate-resistant progression. Progression is defined as any of the following: 1) New lesions or obviously worsening lesions on bone scan within the previous three months; 2) a PSA doubling time of < 3 months; 3) New or progressive symptoms requiring a change in therapy that are referable to the cancer; 4) New extra-osseous lesions within the past 3 months
2. Have progression in the face of a serum testosterone of less than 50 ng/dL, and have either failed or refused chemotherapy
3. Have an Eastern Cooperative Oncology Group (ECOG) performance status 0, 1 or 2
4. Have adequate bone marrow function defined as an absolute peripheral granulocyte count of >/= 1,000/mm^3 and platelet count of >/= 140,000/mm^3; hemoglobin >/= 9.0 g/dL (without transfusion or growth factor support), unless the patient is < 6 weeks from last cancer therapy in which case transfusion is allowed.
5. Have adequate hepatic function defined as a total bilirubin of </= 1.5 mg/dl and AST </= 2* the upper limits of normal
6. Have adequate renal function defined as serum creatinine </= 1.5* the upper limits of normal or creatinine clearance >/= 60 mL/min (measured or calculated). In the absence of hematuria, patients must have either a negative urinalysis for protein (i.e. no more than "trace" by dipstick) or a 24 hour urine collection showing less than 1,000 mg of protein/24 hour. In the presence of hematuria, patients may have up to 2,000 mg of protein/24 hour.
7. Have adequate cardiovascular function as defined by: i) a normal beta-natruetic peptide (BNP) with ii) no signs or symptoms suggestive of cardiac disease and iii) a normal Electrocardiography (ECG). Alternatively, patient not meeting all of these criteria is still eligible if he has both i) an echocardiogram showing an ejection fraction (EF) of 45% or greater (and no more than "mild" diastolic dysfunction) and ii) a Brain Natriuretic Peptide (BNP)of < 200
8. Sign the current Institutional Review Board (IRB) approved informed consent indicating that they are aware of the investigational nature of this study, in keeping with the policies of the institution
9. Age >/= 18 years old

Exclusion Criteria:

1. Small cell prostate cancer
2. Infectious process, which, in the opinion of the investigator, could worsen or its outcome be affected, as a result of the investigational therapy
3. Any of the following in previous 6 months: New York Heart Association (NYHA) Class III/IV congestive heart failure, unstable angina, cerebrovascular accident (including transient ischemic attack), pulmonary embolism or myocardial infarction (by ECG or serologic criteria)
4. Significant co-morbidity that could affect the safety or evaluability of participants, including: a) Chronically uncontrolled hypertension, defined conventionally as consistent systolic pressures above 140 or diastolic pressures above 90 despite therapy. Note that this is NOT a criterion related to particular BP results at the time of assessment for eligibility, nor does it apply to acute BP excursions that are related to iatrogenic causes, acute pain or other transient, reversible causes. (Please see further explanation in the Treatment Plan below)
5. (# 4 cont'd) b) uncontrolled diabetes mellitus (defined as Hgb A1c > 8.5, or symptomatic hypoglycemic episodes > 1 per week during the two months prior to eligibility evaluation, or more than 1 glucose excursion to >300 mg/dL in prior two months--unless clearly iatrogenic and the cause has been eliminated),c) lung disease requiring supplemental oxygen, d) known chronic liver disease, or e) HIV infection
6. Hydronephrosis (either bilateral or involving a solitary kidney) that has not been addressed by means of a nephrostomy or indwelling stent. (Non-obstructive hydronephrosis in setting of prior urinary diversion is allowed.)
7. Overt psychosis, mental disability or being otherwise incompetent to grant informed consent or a history of non-compliance with medical care
8. Patients must not require ongoing therapy with non-steroidal anti-inflammatories (NSAIDs),other than low-dose (i.e. 81 mg or less) aspirin daily, i.v. vancomycin, aminoglycosides, or other potently nephrotoxic drugs, and must agree to abstain from NSAIDs for the duration of their participation in the trial
9. Any other medical condition that in the opinion of the principal investigator would compromise the ability to deliver or evaluate study drug
10. Unwillingness to maintain adequate contraception measures for the entire course of the study
11. Any therapy for prostate cancer (other than ongoing androgen deprivation or associated hormonal therapies such as diethylstilbesterol, low-dose dexamethasone, megace, etc) in the two weeks prior to starting BMTP-11

Min Age: 18 Years | Sex: Male | Healthy Volunteers: No
Age Groups: Adult, Older Adult
Enrollment: 10 (Actual)
Dates: Start 2009-03; Primary Completion 2015-10 (Actual)

PRIMARY OUTCOMES:
Highest tolerable dose of BMTP-11 defined by dose-limiting toxicity | Continuous reassessment, review with weekly dose in 4 week cycle.
  Dose-limiting toxicities defined if they are considered to be possibly, probably or definitely related to study drug:
  • Any grade 3/4 non-hematologic Adverse Event
  • Rise in serum creatinine such that the predicted clearance falls by >40% from baseline
  • Febrile neutropenia
  • Platelet transfusion (either given, or indicated by American Society of Clinical Oncology (ASCO) consensus criteria of 10,000 platelets per microliter)

CONTACTS AND LOCATIONS:
Overall Officials: Christopher Logothetis, MD, Principal Investigator — M.D. Anderson Cancer Center
Locations (1):
- University of Texas MD Anderson Cancer Center, Houston, Texas, United States

REFERENCES:
- [Derived] Pasqualini R, Millikan RE, Christianson DR, Cardo-Vila M, Driessen WH, Giordano RJ, Hajitou A, Hoang AG, Wen S, Barnhart KF, Baze WB, Marcott VD, Hawke DH, Do KA, Navone NM, Efstathiou E, Troncoso P, Lobb RR, Logothetis CJ, Arap W. Targeting the interleukin-11 receptor alpha in metastatic prostate cancer: A first-in-man study. Cancer. 2015 Jul 15;121(14):2411-21. doi: 10.1002/cncr.29344. Epub 2015 Apr 1. PMID 25832466
- See also: University of Texas MD Anderson Cancer Center Website — http://www.mdanderson.org